CLINICAL TRIAL: NCT02610296
Title: A Phase 3, Randomized, Double-blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of QPI-1002 for Prevention of Delayed Graft Function in Recipients of a Donation After Brain Death Older Donor Kidney Transplant
Brief Title: QPI-1002 for Prevention of Delayed Graft Function in Recipients of an Older Donor Kidney Transplant
Acronym: ReGIFT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Quark Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QRK306
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Delayed Graft Function
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- QPI-1002 (Active Comparator): QPI-1002 Injection, single dose
  Interventions: Drug: QPI-1002
- Placebo (Placebo Comparator): isotonic saline
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: QPI-1002 — IV injection
  Arms: QPI-1002
Other: Placebo — isotonic saline
  Arms: Placebo

SUMMARY:
The purpose of this trial is to evaluate the reduction in incidence and severity of delayed graft function with kidney allografts from donors >45 years after brain death (DBD).

DETAILED DESCRIPTION:
This is a Phase 3 randomized, placebo-controlled, double-blind, multi-center trial stratified by donor age and by region to evaluate the reduction in incidence and severity of delayed graft function with kidney allografts from DBD donors who were at least 45 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Has the ability to understand the requirements of the study, is able to provide written informed consent and is willing and able to comply with the requirements of the study protocol.
* Male or female at least 18 years of age.
* Has dialysis dependent renal failure initiated at least 2 months prior to transplantation.
* Is to be a recipient of a transplant from a deceased donor (brain death criteria) ≥ 45 years of age.
* Based on donor age, the following requirements for the risk of DGF (determined using the Irish DGF risk assessment nomogram) and cold ischemia time (CIT) must be met:

  * Donor age 45 - 59 years: estimated DGF risk ≥ 20% and estimated CIT ≥ 10 hour
  * Donor age ≥ 60 years: no minimum estimated DGF risk or minimum estimated CIT
* Is able to comply with the requirement of antibody induction therapy with rabbit polyclonal anti-thymocyte globulin or anti-CD25 (anti-IL2R) monoclonal antibodies per center standard of care.
* Must be up-to-date on cancer screening according to site-specific guidelines and past medical history must be negative for biopsy-confirmed malignancy within 5 years of randomization, with the exception of adequately treated basal cell or squamous cell carcinoma in situ or carcinoma of the cervix in situ.

Exclusion Criteria:

* Recipient of a live donor kidney or a kidney from a donation after cardiac death (DCD) donor.
* Recipient of donor kidney preserved with normothermic machine perfusion.
* Scheduled to undergo multiorgan transplantation.
* Has a planned transplant of kidneys that are implanted en bloc (dual kidney transplant).
* Has planned transplant of dual kidneys (from the same donor) transplanted not en bloc.
* Has lost first kidney transplant due to graft thrombosis.
* Is scheduled for transplantation of a kidney from a donor who is known to have received an investigational therapy under another IND/CTA for ischemic/reperfusion injury immediately prior to organ recovery.
* Is scheduled to receive an ABO-incompatible donor kidney.
* Has a positive T- or B-cell cross-match by NIH anti-globulin lymphocytotoxicity method or CDC crossmatch method, if performed.
* Has a positive T- or B-cell flow cross-match AND donor specific anti-HLA antibody (DSA) detected by flow cytometry, Luminex® based antigen-specific anti-HLA antibody testing, or by similar methodology, if performed.
* Has undergone desensitization to remove donor specific anti-HLA antibodies prior to transplantation.
* Has participated in an investigational study within the last 30 days or received an investigational product within 5 half-lives of the study drug administration, whichever is longest.
* Has known allergy to or has participated in a prior study with siRNA.
* Has a history of HBV (Note: subjects with a serological profile suggestive of clearance, or prior antiviral treatment of a prior HBV infection, may be enrolled with the approval of the Medical Monitor).
* Has a history of HIV.
* Recipient of a known HIV positive donor kidney.
* Is HCV-positive (detectable HCV RNA) (Note: Subjects at least 24 weeks from completion of treatment with an approved antiviral regimen and who remain free of HCV as determined by HCV RNA testing may be enrolled. Subjects who have been cleared of HCV virus after treatment with an unapproved regimen should be approved by the Medical Monitor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
The number of dialysis sessions through Day 30 for subjects who started dialysis beginning in the first 7 days post-transplant. | Day 0 to Day 30

SECONDARY OUTCOMES:
The proportion of subjects requiring dialysis for any reason in the first 7 days post-transplant. | Day 0 to Day 7
The proportion of subjects with a decrease in serum creatinine of ≥ 10% on three consecutive days in the first 7 days post-transplant. | Day 0 to Day 7

CONTACTS AND LOCATIONS:
Overall Officials: John Holman, M.D.,Ph.D., Study Director — Quark Pharmaceuticals
Locations (84):
- United States (36):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado, Denver, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Georgetown Transplant Institute, Washington D.C., District of Columbia
  - University of Florida Health, Shands Hospital, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Louisville, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Erie County Medical Center, Buffalo, New York
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Columbia University, New York, New York
  - New York - Presbyterian Hospital / Weill Cornell Medical Center, New York, New York
  - SUNY Upstate NY University Hospital, Syracuse, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Integris Nazih Zuhdi Transplant Institute, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - Baylor All Saints, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Argentina (2):
  - Hospital Universitario Austral, Buenos Aires
  - Instituto de Nefrología Trasplante Renal y Renopancreatico, Buenos Aires
- Australia (5):
  - John Hunter Hospital, New Lambton, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide, Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
- Belgium (2):
  - UZ Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier - Universitaire de Liège, Liège
- Brazil (7):
  - Hospital Geral de Fortaleza, Fortaleza, Ceará
  - Instituto de Medicina Integral Prof. Fernando Figueira (IMIP), Recife, Pernambuco
  - Hospital São Francisco de Assis, Rio de Janeiro, Rio de Janeiro
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Fundação Oswaldo Ramos - Hospital do Rim, São Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
- Canada (4):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - St. Michael's Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Klinika nefrologie IKEM, Prague, Czechia
- France (7):
  - Hôpital Pellegrin, Bordeaux
  - Hospital Henri Mondor - Créteil, Créteil
  - Centre Hospitalier Universitaire de Grenoble, La Tronche
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Pasteur, Nice
  - Hôpital Necker, Paris
  - Centre Hospitalier Universitaire de Rangueil, Toulouse
- Germany (8):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Charité - Universitätsmedizin Berlin, Campus Virchow-Klinikum (CVK), Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Klinik für Nieren und Hochdruckerkrankungen, Hanover
  - University Hospital Schleswig Holstein, Campus Kiel, Kiel
  - Universitätsklinikum Tübingen, Tübingen
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Leids Universitair Medisch Centrum, Leiden
  - Maastricht University Medical Centre, Maastricht
- Spain (9):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d´Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza